CLINICAL TRIAL: NCT05718869
Title: A Phase 2 Study With a Safety Lead-In of the Anti-CD19 Antibody Tafasitamab With the BTK Inhibitor Zanubrutinib in Newly Diagnosed Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL) - TaZa CLL Study
Brief Title: Tafasitamab and Zanubrutinib for the Treatment of Patients With Newly Diagnosed Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma, TaZA CLL Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22183; NCI-2022-10205 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22183 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-01-20; First posted 2023-02-08 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Specimen Handling; Biopsy; tafasitamab; Immunoglobulins; Disulfides; zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (tafasitamab and zanubrutinib) (Experimental): Patients receive tafasitamab IV and zanubrutinib PO on study. Patients also undergo collection of blood samples on study and undergo CT scan and bone marrow biopsy throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Biological: Tafasitamab; Drug: Zanubrutinib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Biological: Tafasitamab — Given IV
  Other Names: Immunoglobulin, Anti-(Human Cd19 Antigen) (Human-mus musculus Monoclonal MOR00208 Heavy Chain), Disulfide with Human-mus musculus Monoclonal MOR00208 .Kappa.-chain, Dimer; Monjuvi; MOR-00208; MOR00208; MOR208; Tafasitamab-cxix; XmAb5574
Drug: Zanubrutinib — Given PO
  Other Names: BGB-3111; Brukinsa; BTK-InhB

SUMMARY:
This phase II trial tests how well tafasitamab and zanubrutinib works in treating patients with newly diagnosed chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL). Tafasitamab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Zanubrutinib is in a class of medications called kinase inhibitors. It works by blocking the action of a protein that signals cancer cells to multiply. This may stop the growth and spread of cancer cells. Giving tafasitamab and zanubrutinib in combination may kill more cancer cells in patients with CLL/SLL than giving either treatment alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety/tolerability of tafasitamab and zanubrutinib (as assessed by unacceptable toxicity) in patients with newly diagnosed CLL. (Safety lead-in) II. To evaluate the anti-tumor activity of tafasitamab and zanubrutinib as assessed by complete response (CR) rate per International Workshop on CLL (iwCLL) 2018 criteria in patients with newly diagnosed CLL. (Phase 2)

SECONDARY OBJECTIVES:

I. To assess the toxicity of the combination of tafasitamab and zanubrutinib through evaluation of toxicities.

II. To obtain estimates of overall response rate (ORR), progression-free survival (PFS), and duration of response (DOR).

III. To assess the undetectable minimal residual disease (uMRD) rate in response to tafasitamab and zanubrutinib.

EXPLORATORY OBJECTIVES:

I. To assess the effect of tafasitamab and zanubrutinib combination on immune function of T cells and NK cells.

II. To explore mechanisms of resistance to the combination of tafasitamab and zanubrutinib.

III. To investigate the association of established biomarkers (chromosomal abnormalities, immunoglobulin heavy chain [IGHV] mutational status, TP53 mutational status) with response (ORR and PFS) to tafasitamab and zanubrutinib in patients with CLL.

OUTLINE: This is a dose-escalation study of zanubrutinib followed by a phase II study.

Patients receive tafasitamab intravenously (IV) and zanubrutinib orally (PO) on study. Patients also collection of blood samples on study and undergo computed tomography (CT) scan and bone marrow biopsy throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Age: >= 18 years
* Eastern Cooperative Oncology Group (ECOG) =< 2
* Histologically or flow cytometry confirmed diagnosis of B-CLL/SLL as documented by medical records and with histology based on criteria established by the World Health Organization (WHO)
* No prior treatment for CLL, except steroids and/or rituximab to treat autoimmune complications
* Active disease meeting criteria for requiring treatment per the iwCLL 2018 guidelines

  * A minimum of any one of the following constitutional symptoms:

    * Unintentional weight loss > 10% within the previous 6 months prior to screening
    * Extreme fatigue (unable to work or perform usual activities)
    * Fevers of greater than 100.5 degrees Fahrenheit (F) for >= 2 weeks without evidence of infection
    * Night sweats without evidence of infection
  * Evidence of progressive marrow failure as manifested by the development of, or worsening of anemia or thrombocytopenia
  * Massive (i.e., > 6 cm below the left costal margin), progressive or symptomatic splenomegaly
  * Massive nodes or clusters (i.e., > 10 cm in longest diameter) or progressive lymphadenopathy
  * Progressive lymphocytosis with an increase of > 50% over a 2-month period, or an anticipated doubling time of less than 6 months
  * Autoimmune anemia or thrombocytopenia that is poorly responsive to corticosteroids
  * Symptomatic or functional extranodal involvement (eg, skin, kidney, lung, spine)
* Participant must be able to swallow tablets or capsules. A participant with any gastrointestinal disease that would impair ability to swallow, retain, or absorb drug is not eligible
* Absolute neutrophil count (ANC) >= 1,000/mm^3 unless due to bone marrow involvement

  * NOTE: Growth factor is not permitted within 14 days of ANC assessment unless cytopenia is secondary to disease involvement
* Platelets >= 75,000/mm^3 unless due to bone marrow involvement, and independent of transfusion support, with no active bleeding
* Direct bilirubin =< 1.5 X upper limit of normal (ULN) (unless has Gilbert's disease or compensated hemolysis directly attributable to CLL)
* Aspartate aminotransferase (AST) =< 2.5 X ULN
* Alanine aminotransferase (ALT) =< 2.5 X ULN
* Estimated creatinine clearance of >= 30 mL/min using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula
* IF NOT RECEIVING ANTICOAGULANTS: International normalized ratio (INR) OR prothrombin (PT) =< 1.5 x ULN; IF ON ANTICOAGULANT THERAPY: PT must be within therapeutic range of intended use of anticoagulants
* IF NOT RECEIVING ANTICOAGULANTS: Activated partial thromboplastin time (aPTT) =< 1.5 x ULN; IF ON ANTICOAGULANT THERAPY: aPTT must be within therapeutic range of intended use of anticoagulants
* Women of childbearing potential (WOCBP): negative serum pregnancy test
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 3 months after the last dose of protocol therapy

  * A woman is considered of childbearing potential, ie, fertile, following menarche and until becoming postmenopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy. Contraception methods include the following:

    * Combined (estrogen- and progestogen- containing) hormonal contraception associated with the inhibition of ovulation or oral, intravaginal, or transdermal
    * Progestogen-only hormonal contraception associated with the inhibition of ovulation or oral, injectable, implantable
    * An intrauterine device
    * Intrauterine hormone-releasing system
    * Bilateral tubal occlusion vasectomized partner (provided that the vasectomized partner is the sole sexual partner of the woman of childbearing potential study participant and that the vasectomized partner has received medical assessment of surgical success)
    * Sexual abstinence (defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatment, starting the day prior to first dose of study drug, for the duration of the study, and for >= 90 days after the last dose of zanubrutinib or ibrutinib. Total sexual abstinence should only be used as a contraceptive method if it is in line with the patients' usual and preferred lifestyle. Periodic abstinence (eg, calendar, ovulation, symptothermal, postovulation methods), declaration of abstinence for the duration of exposure to investigational medicinal product, and withdrawal are not acceptable methods of contraception. Of note, barrier contraception (including male and female condoms with or without spermicide) is not considered a highly effective method of contraception, and, if used, this method must be used in combination with another acceptable method listed above. If patient is using hormonal contraceptives such as birth control pills or devices, a barrier method of contraception (eg, condoms) must also be used. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle-stimulating hormone level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single follicle-stimulating hormone measurement is insufficient

Exclusion Criteria:

* Chronic use of corticosteroids in excess of 20 mg/day prednisone or its equivalent
* Major surgery (under general anesthesia) within 30 days prior to therapy
* Uncontrolled coagulopathy or bleeding disorder. Direct oral anticoagulants are allowed
* Use of moderate or strong cytochrome P450 3A4 (CYP3A4) inducer within 2 weeks of the first day of study therapy. CYP3A inhibitors are allowed.

  * For patients intended to enroll on dose level (DL) -1 use of strong CYP3A inhibitors will be prohibited on-therapy and their use must be stopped at minimum 2 weeks prior to the first day of study therapy
* Exposure to vaccination with live vaccine within 30 days prior to cycle 1 day 1 (C1D1), or anticipated need for such vaccination during treatment
* History of prior malignancy except:

  * Malignancy treated with curative intent and no known active disease present for >= 2 years prior to initiation of therapy on current study
  * Adequately treated non-melanoma skin cancer or lentigo maligna (melanoma in situ) without evidence of disease
  * Adequately treated in situ carcinomas (e.g., cervical, esophageal, etc.) without evidence of disease
  * Asymptomatic prostate cancer managed with "watch and wait" strategy
* Uncontrolled immune hemolysis or thrombocytopenia (positive direct antiglobulin test in absence of hemolysis or history of immune-mediated cytopenias are not exclusions)
* Known positive test result for SARS-CoV-2 unless follow-up test was negative or investigator deems the infection is fully resolved
* Known positive test result for hepatitis C (hepatitis C virus [HCV] antibody serology testing) and a positive test result for HCV ribonucleic acid (RNA). Participants with positive serology are eligible in case of negative HCV RNA test results
* Known positive test result for chronic hepatitis B virus (HBV) infection (defined by hepatitis B virus surface antigen [HBsAg] positivity)

  * Participants with occult or prior HBV infection (defined as negative HBsAg and positive total hepatitis B core antibody) may be included if HBV deoxyribonucleic acid (DNA) was undetectable, provided that they are willing to undergo ongoing DNA testing.
  * Antiviral prophylaxis may be administered as per institutional guidelines.
  * Participants who have protective titers of HBsAb after vaccination or prior but cured hepatitis B are eligible
* Known seropositive for or history of active viral infection with human immunodeficiency virus (HIV)
* Clinically significant cardiovascular disease including the following:

  * Myocardial infarction within 6 months before screening
  * Unstable angina within 3 months before screening
  * New York Heart Association class III or IV congestive heart failure
  * History of clinically significant arrhythmias (eg, sustained ventricular tachycardia, ventricular fibrillation, Torsades de Pointes)
  * QTcF > 480 milliseconds based on Fridericia's formula
  * History of Mobitz II second-degree or third-degree heart block without a permanent pacemaker in place
* Known severe chronic obstructive pulmonary disease (COPD)
* Known hepatic cirrhosis or severe pre-existing hepatic impairment
* Major surgery (requiring general anesthesia) within 14 days before the first dose of study drug or a scheduled surgery during study period
* Patients with clinically significant medical condition of malabsorption, inflammatory bowel disease, chronic conditions which manifest with diarrhea, refractory nausea, vomiting or any other condition that will interfere significantly with drug absorption
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-05-18 (Actual); Primary Completion 2026-04-19 (Estimated); Study Completion 2026-04-19 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) rate | Up to 5 years
  Defined as the proportion of response evaluable patients who achieve a complete response according to International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2018 guidelines on study before any documented disease progression or any subsequent chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL) treatment. CR rate will be estimated by the proportion of response-evaluable patients achieving CR, along with the 95% exact binomial confidence interval.
Incidence of adverse events | Up to 5 years
  Grading of toxicities will be according to National Cancer Institute's Common Terminology Criteria for Adverse Events version 5. Observed toxicities will be summarized by type (organ affected or laboratory determination such as absolute neutrophil count), severity, and attribution.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 5 years
  Defined as the proportion of response evaluable patients who achieve complete response or partial response (PR) according to iwCLL 2018 guidelines on study before any documented disease progression or any subsequent CLL/SLL treatment. ORR will be estimated similar to CR rate.
Progression-free survival (PFS) | From start of protocol treatment to disease relapse/progression or death due to any cause, assessed up to 5 years
  PFS will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% confidence interval will be constructed based on log-log transformation. Median PFS will be estimated when available.
Duration of response (DOR) | From the first achievement of CR or PR to disease progression/relapse or death due to any cause, assessed up to 5 years
  DOR will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% confidence interval will be constructed based on log-log transformation. Median DOR will be estimated when available.
Undetectable minimal residual disease (uMRD) rate | On day 1 of cycles 1, 4, 7, 13, 18, and 24 ( each cycle is 28 days)
  Defined as the proportion of patients who achieve uMRD status, defined as < 10^-4 CLL cells by clonoSEQ, among those tested for minimal residual disease.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Mei, Principal Investigator — City of Hope Medical Center
Locations (3):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida